CLINICAL TRIAL: NCT07137754
Title: Effect and Cost-effectiveness of a Physiotherapy-led Care Model for Patients Referred to an Emergency Department Due to Musculoskeletal Injuries: A Multicentre Quasi-randomized Clinical Trial
Brief Title: Effect and Cost of a Physiotherapy-led Care Model in Emergency Departments for Patients With Minor Musculoskeletal Injuries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Slagelse Hospital (Other); Gødstrup Hospital (Other); Université de Montréal (Other); Independent Research Fund Denmark (Industry); University of Aarhus (Other); Danske Fysioterapeuter (Other)
Responsible Party: Principal Investigator, Nanna Rolving, Associate professor, Aarhus University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Journal no. 1-10-72-137-24; 4285-00270B (Other Grant/Funding Number: Independent Research Fund Denmark)
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Musculoskeletal Disorders; Emergency Care; Physiotherapy
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced practice physiotherapy (Experimental): Advanced practice physiotherapists will independently diagnose, manage and discharge patients
  Interventions: Other: Advanced practice physiotherapy
- Usual care (Active Comparator): Nurses and physicians in the emergency department will diagnose, manage and discharge patients as per usual care
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Advanced practice physiotherapy — Physiotherapists undergoing post-graduate education as advanced practice physiotherapists will independently diagnose, manage and discharge patients.
  Arms: Advanced practice physiotherapy
Other: Usual Care — Nurses and physicians in the emergency department will diagnose, manage and discharge patients as usual
  Arms: Usual care

SUMMARY:
Both in Denmark and internationally, emergency departments have been overwhelmed for several years by a growing number of patients, combined with a shortage of doctors and nurses. This problem is expected to continue because the number of elderly people with multiple health problems is increasing. To keep providing good quality care in emergency departments, we need to consider new ways of organizing treatment.

In Canada, Australia, and the UK, some hospitals have tried a model where specially trained physiotherapists examine and treat patients who come in with muscle and joint injuries and pain. Since these patients make up about 25% of all those referred to emergency departments, this model could help take some pressure off doctors and nurses. That way, doctors and nurses can spend more time caring for seriously ill patients who need urgent help.

Several studies on these physiotherapist-led models show benefits for both patients and the healthcare system. Patients report being more satisfied and better informed about their injury and treatment. They wait less, have fewer unnecessary tests, and need fewer repeat visits to the emergency department.

However, similar studies have never been done in Scandinavia, even though some Danish emergency departments have tested similar models. Healthcare systems and the education of physiotherapists differ between Scandinavian countries and the countries mentioned above. So, we don't know if we would see the same benefits here. Also, there has been no research on whether this model is cost-effective, which is important for decision-makers when planning future healthcare budgets.

With this research project, we want to test a model in Danish hospitals where specially trained physiotherapists take care of examining, treating, and discharging patients with muscle and joint pain and injuries. We will look at how this model affects patient experiences (like pain and satisfaction) and clinical outcomes (like repeat emergency visits and use of imaging tests), compared to the usual practice where doctors handle these patients. We will also study whether the model is cost-effective, meaning whether the benefits of using this approach are worth the costs, or even greater than the costs.

The study will be conducted at 4-5 hospitals, where a total of 800 patients with minor musculoskeletal injuries will be included in connection with their visit at the emergency department. Patients will receive questionnaires at 1, 4, 12 and 26 weeks after injury regarding patient reported outcomes. Register data will be retrieved at 26 weeks regarding the patients' health care use during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Musculoskeletal pain and injury to the upper or lower extremities
* Triaged non-urgent (blue) in the emergency department
* Speaks and understands Danish

Exclusion Criteria:

* High velocity trauma
* Cognitively unable to participate
* Non-malignant conditions (cancer, inflammation, infection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Brief pain inventory short form | From baseline (time of injury) to 12 weeks follow-up
  BPI short form is a self-reported questionnaire, using the 7 items pain interference on functional ability, mood, sleep and work. The patient completes the assessment at baseline, 1, 4, 12 and 26 weeks after injury
Euroqol 5 Dimensions 5 Levels | From baseline to 26 weeks
  The EQ5D assesses health-related quality of life using 5 items. It is used as the primary outcome for qualculation of QUALYs in the health economic analysis.

SECONDARY OUTCOMES:
Visit-specific satisfaction questionnaire | Is collected at week 1 after baseline
  VSQ-9 is a selfreported questionnaire with 9 items on different aspects of patient satisfaction with their visit to the emergency department
PROMIS short form physical function | From baseline to 12 weeks after.
  The questionnaire contains 8 questions on limitations in functional ability due to injuries in the lowe extremeties. It is collected via self-reported questionnaires at baseline, weeks 1, 4, 12 and 26 after baseline
PROMIS short form upper extremety | From baseline to 12 weeks
  Contains questions about functional limitations due to injuries in the upper extremeties. Measured at baseline, weeks 1, 4, 12 and 26 after discharge
Work Productivity and Activity Impairment | From baseline to 12 weeks
  The WPAI measures number of hours missed from work, volunteer work (unpaid work) and studies due to health related issues. Further it measures hours with reduced productivity at work due to health related issues. Assessed at baseline, weeks 1, 4, 12 and 26 using self-reported questionnaires
Return-visits to emergency department | From baseline to 12 week follow-up
  Return-visits and phone calls to the emergency department due to the same injury during follow-up, assessed using self-report and register-based data.
Health care use in primary care | From baseline to 26 week follow-up
  Includes visits with general practice and physiotherapy practice during follow-up. This will be collected via the National Health Service Register

CONTACTS AND LOCATIONS:
Overall Officials: Nanna Rolving, Associate professor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Decision on IPD sharing plan awaits steering group meeting, with the expectation that a plan for IPD sharing will be registered later on.